CLINICAL TRIAL: NCT00042705
Title: Asthma Severity in Children and Environmental Agents
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 5410-CP-001
Record Dates: First submitted 2002-08-05; First posted 2002-08-06 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: asthma; indoor allergens
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study measures residential exposures (indoor allergens, mold, nitrogen dioxide, nicotine) and relates exposure levels to daily symptoms (wheeze, persistent cough, chest tightness, shortness of breath) and medication use, in a population of children with physician diagnosed asthma, followed for 12 months.

ELIGIBILITY:
* Siblings of a birth cohort recruited 1997-1999
* Age less than 11 years
* Physician diagnosed asthma
* Active symptoms (wheeze, persistent cough, chest tightness, shortness of breath) or medication use in the 12 months prior to enrollment.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2000-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Center for Perinatal, Pediatric & Environmental Epidemiology, New Haven, Connecticut, United States